CLINICAL TRIAL: NCT04882371
Title: Comparison of MRI With PET / CT in the Evaluation of Response to Neoadjuvant Therapy Based on the Molecular Subtypes of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Cem Ilgin Erol (Other)
Responsible Party: Sponsor-Investigator, Cem Ilgin Erol, MD, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Other Study IDs: 2020-0327
Record Dates: First submitted 2021-05-08; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Chemotherapy Effect
Keywords: Breast Neoplasms; Neoadjuvant chemotherapy; RECIST; PERCIST
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Magnetic Resonance Imaging; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI RECIST: Radiological responses were evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) and changes in contrast enhancement patterns on MRI
  Interventions: Drug: Chemotherapy; Diagnostic Test: Magnetic Resonance Imaging (MRI)
- PET-CT PERCIST: Radiological responses were evaluated according to the classification of PET Response Criteria in Solid Tumors (PERCIST) on PET-CT.
  Interventions: Drug: Chemotherapy; Diagnostic Test: Positron emission tomography - Copmputer Tomography (PET-CT)

INTERVENTIONS:
Drug: Chemotherapy — Neoadjuvant Chemotherapy for Breast Cancer
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Performed contrasted MRI for evaluate response of neoadjuvant chemotherapy
  Groups: MRI RECIST
Diagnostic Test: Positron emission tomography - Copmputer Tomography (PET-CT) — Performed contrasted PET-CT for evaluate response of neoadjuvant chemotherapy
  Groups: PET-CT PERCIST

SUMMARY:
The current study aims to determine the diagnostic accuracy of Magnetic Resonance Imaging (MRI) and Positron Emission Tomography- Computed Tomography (PET-CT) in predicting a pathological response of molecular subtypes of breast cancer to neoadjuvant chemotherapy (NAC).

DETAILED DESCRIPTION:
Eighty-eight patients with breast cancer who had undergone surgery after NAC were retrospectively analyzed between January 2018 and May 2020, at the general surgery clinic of Istanbul Medeniyet University Göztepe Training and Research Hospital. Demographic data, clinical findings, tumor markers, radiologic findings and pathology data were documented. With the use of MRI and / or PET-CT obtained before and after NAC, tumor staging was performed, and tumor size and the presence of metastatic lymph nodes and radiological response to NAC were evaluated. The response to NAC was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST) and contrast enhancement patterns described by Tozaki et al. on MRI, and the classification PET Response Criteria in Solid Tumors (PERCIST) on PET-CT. The postoperative pathology study reported the followings: the size and histopathologic type of the tumor, its hormone receptor status, staining intensities (Allred score), HER-2 positivity, Ki-67 proliferation percentages, and the molecular subtypes; the presence and number of metastatic lymph nodes, the response of the tumor and, the metastatic lymph node, if any, to NAC according to the Sataloff classification. Patients with a Sataloff score of "A" were considered to have a pCR, those with the scores of "B" or "C" were considered to have a partial response. When examining the Sataloff scores, the presence of pCR in both the primary tumor and axilla was evaluated and compared with the presence of radiological complete response on MRI and / or PET-CT. In addition, the sensitivities of MRI and PET-CT in predicting pCR in patients undergoing NAC were statistically compared based on the molecular subtypes. Patients whose MRI and PET-CT findings were consistent with histopathologic data were included in the "Radiology-Pathology agreement " group. The sensitivity of imaging methods was determined by examining the rates of agreement in the molecular subgroups. The Statistical Package for Social Sciences software for Windows version 20 (SPSS Inc.; Chicago, IL, USA) was used for all analyses. Normality was assessed by the Shapiro-Wilk test. Categorical variables were compared using chi-square or, where appropriate, Fisher's exact test. The Mc-Nemar test was used for paired categorical data. Trends in tables larger than 2x2 were examined with the linear-by-linear association test. Kruskal-Wallis test was used to compare non-normal distributed variables in three groups. Cohen's kappa (κ) was calculated to test the agreement between the classifications of radiology and pathology.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* Breast cancer patients
* Had neoadjuvant chemotherapy before surgery
* Had undergone surgery after chemotherapy

Exclusion Criteria:

* Younger than 18
* History of surgery for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer who had undergone surgery after neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Radiological evaluation of response to neoadjuvant chemotheraphy for breast cancer | 2 months
  All patient had neoadjuvant chemotherapy, then a group of patient evaluated with MRI and the other group of patient with PET-CT

SECONDARY OUTCOMES:
Pathological evaluation of response to neoadjuvant chemotheraphy for breast cancer | 2 months
  Surgery was performed for all patient after neoadjuvant chemotherapy. Pathological datas were analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Goztepe City Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization, Fact Sheets, Detail, Cancer. https://www.who.int/news-room/fact-sheets/detail/cancer
- [Background] International Agency for Research on Cancer, Globocan 2018 Report. https://www.uicc.org/news/global-cancer-data-globocan-2018
- [Background] Gianni L, Eiermann W, Semiglazov V, Lluch A, Tjulandin S, Zambetti M, Moliterni A, Vazquez F, Byakhov MJ, Lichinitser M, Climent MA, Ciruelos E, Ojeda B, Mansutti M, Bozhok A, Magazzu D, Heinzmann D, Steinseifer J, Valagussa P, Baselga J. Neoadjuvant and adjuvant trastuzumab in patients with HER2-positive locally advanced breast cancer (NOAH): follow-up of a randomised controlled superiority trial with a parallel HER2-negative cohort. Lancet Oncol. 2014 May;15(6):640-7. doi: 10.1016/S1470-2045(14)70080-4. Epub 2014 Mar 20. PMID 24657003
- [Background] Cardoso F, Costa A, Norton L, Senkus E, Aapro M, Andre F, Barrios CH, Bergh J, Biganzoli L, Blackwell KL, Cardoso MJ, Cufer T, El Saghir N, Fallowfield L, Fenech D, Francis P, Gelmon K, Giordano SH, Gligorov J, Goldhirsch A, Harbeck N, Houssami N, Hudis C, Kaufman B, Krop I, Kyriakides S, Lin UN, Mayer M, Merjaver SD, Nordstrom EB, Pagani O, Partridge A, Penault-Llorca F, Piccart MJ, Rugo H, Sledge G, Thomssen C, Van't Veer L, Vorobiof D, Vrieling C, West N, Xu B, Winer E; European School of Oncology; European Society of Medical Oncology. ESO-ESMO 2nd international consensus guidelines for advanced breast cancer (ABC2). Breast. 2014 Oct;23(5):489-502. doi: 10.1016/j.breast.2014.08.009. Epub 2014 Sep 20. No abstract available. PMID 25244983
- [Background] Cortazar P, Zhang L, Untch M, Mehta K, Costantino JP, Wolmark N, Bonnefoi H, Cameron D, Gianni L, Valagussa P, Swain SM, Prowell T, Loibl S, Wickerham DL, Bogaerts J, Baselga J, Perou C, Blumenthal G, Blohmer J, Mamounas EP, Bergh J, Semiglazov V, Justice R, Eidtmann H, Paik S, Piccart M, Sridhara R, Fasching PA, Slaets L, Tang S, Gerber B, Geyer CE Jr, Pazdur R, Ditsch N, Rastogi P, Eiermann W, von Minckwitz G. Pathological complete response and long-term clinical benefit in breast cancer: the CTNeoBC pooled analysis. Lancet. 2014 Jul 12;384(9938):164-72. doi: 10.1016/S0140-6736(13)62422-8. Epub 2014 Feb 14. PMID 24529560
- [Background] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986
- [Background] Abedi M, Farrokh D, Shandiz Homaei F, Joulaee A, Anbiaee R, Zandi B, Gity M, Sayah HR, Abedi MS. The validity of MRI in evaluation of tumor response to neoadjuvant chemotherapy in locally advanced breast cancer. Iran J Cancer Prev. 2013 Winter;6(1):28-35. PMID 25250107
- [Background] Gonzalez-Angulo AM, Morales-Vasquez F, Hortobagyi GN. Overview of resistance to systemic therapy in patients with breast cancer. Adv Exp Med Biol. 2007;608:1-22. doi: 10.1007/978-0-387-74039-3_1. PMID 17993229
- [Background] Wang H, Mao X. Evaluation of the Efficacy of Neoadjuvant Chemotherapy for Breast Cancer. Drug Des Devel Ther. 2020 Jun 18;14:2423-2433. doi: 10.2147/DDDT.S253961. eCollection 2020. PMID 32606609
- [Background] Dhillon GS, Bell N, Ginat DT, Levit A, Destounis S, O'Connell A. Breast MR Imaging: What the Radiologist Needs to Know. J Clin Imaging Sci. 2011;1:48. doi: 10.4103/2156-7514.85655. Epub 2011 Oct 3. PMID 22059150
- [Background] Nunes LW, Schnall MD, Orel SG, Hochman MG, Langlotz CP, Reynolds CA, Torosian MH. Correlation of lesion appearance and histologic findings for the nodes of a breast MR imaging interpretation model. Radiographics. 1999 Jan-Feb;19(1):79-92. doi: 10.1148/radiographics.19.1.g99ja0379. PMID 9925393
- [Background] Rausch DR, Hendrick RE. How to optimize clinical breast MR imaging practices and techniques on Your 1.5-T system. Radiographics. 2006 Sep-Oct;26(5):1469-84. doi: 10.1148/rg.265055176. PMID 16973776
- [Background] Tozaki M, Kobayashi T, Uno S, Aiba K, Takeyama H, Shioya H, Tabei I, Toriumi Y, Suzuki M, Fukuda K. Breast-conserving surgery after chemotherapy: value of MDCT for determining tumor distribution and shrinkage pattern. AJR Am J Roentgenol. 2006 Feb;186(2):431-9. doi: 10.2214/ajr.04.1520. PMID 16423949
- [Background] Kim TH, Kang DK, Yim H, Jung YS, Kim KS, Kang SY. Magnetic resonance imaging patterns of tumor regression after neoadjuvant chemotherapy in breast cancer patients: correlation with pathological response grading system based on tumor cellularity. J Comput Assist Tomogr. 2012 Mar-Apr;36(2):200-6. doi: 10.1097/RCT.0b013e318246abf3. PMID 22446360
- [Background] Hegarty C, Collins CD. PET/CT and breast cancer. Cancer Imaging. 2010 Oct 4;10 Spec no A(1A):S59-62. doi: 10.1102/1470-7330.2010.9031. PMID 20880780
- [Background] Park SH, Moon WK, Cho N, Chang JM, Im SA, Park IA, Kang KW, Han W, Noh DY. Comparison of diffusion-weighted MR imaging and FDG PET/CT to predict pathological complete response to neoadjuvant chemotherapy in patients with breast cancer. Eur Radiol. 2012 Jan;22(1):18-25. doi: 10.1007/s00330-011-2236-x. Epub 2011 Aug 16. PMID 21845462
- [Background] Basu S, Chen W, Tchou J, Mavi A, Cermik T, Czerniecki B, Schnall M, Alavi A. Comparison of triple-negative and estrogen receptor-positive/progesterone receptor-positive/HER2-negative breast carcinoma using quantitative fluorine-18 fluorodeoxyglucose/positron emission tomography imaging parameters: a potentially useful method for disease characterization. Cancer. 2008 Mar 1;112(5):995-1000. doi: 10.1002/cncr.23226. PMID 18098228
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Mauri D, Pavlidis N, Ioannidis JP. Neoadjuvant versus adjuvant systemic treatment in breast cancer: a meta-analysis. J Natl Cancer Inst. 2005 Feb 2;97(3):188-94. doi: 10.1093/jnci/dji021. PMID 15687361
- [Background] Spring LM, Fell G, Arfe A, Sharma C, Greenup R, Reynolds KL, Smith BL, Alexander B, Moy B, Isakoff SJ, Parmigiani G, Trippa L, Bardia A. Pathologic Complete Response after Neoadjuvant Chemotherapy and Impact on Breast Cancer Recurrence and Survival: A Comprehensive Meta-analysis. Clin Cancer Res. 2020 Jun 15;26(12):2838-2848. doi: 10.1158/1078-0432.CCR-19-3492. Epub 2020 Feb 11. PMID 32046998
- [Background] Boughey JC, McCall LM, Ballman KV, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Flippo-Morton T, Hunt KK. Tumor biology correlates with rates of breast-conserving surgery and pathologic complete response after neoadjuvant chemotherapy for breast cancer: findings from the ACOSOG Z1071 (Alliance) Prospective Multicenter Clinical Trial. Ann Surg. 2014 Oct;260(4):608-14; discussion 614-6. doi: 10.1097/SLA.0000000000000924. PMID 25203877
- [Background] Resende U, Cabello C, Oliveira Botelho Ramalho S, Zeferino LC. Predictors of Pathological Complete Response in Women with Clinical Complete Response to Neoadjuvant Chemotherapy in Breast Carcinoma. Oncology. 2018;95(4):229-238. doi: 10.1159/000489785. Epub 2018 Jul 19. PMID 30025385
- [Background] Tang S, Xiang C, Yang Q. The diagnostic performance of CESM and CE-MRI in evaluating the pathological response to neoadjuvant therapy in breast cancer: a systematic review and meta-analysis. Br J Radiol. 2020 Aug;93(1112):20200301. doi: 10.1259/bjr.20200301. Epub 2020 Jul 2. PMID 32574075
- [Background] Tateishi U, Miyake M, Nagaoka T, Terauchi T, Kubota K, Kinoshita T, Daisaki H, Macapinlac HA. Neoadjuvant chemotherapy in breast cancer: prediction of pathologic response with PET/CT and dynamic contrast-enhanced MR imaging--prospective assessment. Radiology. 2012 Apr;263(1):53-63. doi: 10.1148/radiol.12111177. PMID 22438441
- [Background] Jones EF, Hathi DK, Freimanis R, Mukhtar RA, Chien AJ, Esserman LJ, Van't Veer LJ, Joe BN, Hylton NM. Current Landscape of Breast Cancer Imaging and Potential Quantitative Imaging Markers of Response in ER-Positive Breast Cancers Treated with Neoadjuvant Therapy. Cancers (Basel). 2020 Jun 9;12(6):1511. doi: 10.3390/cancers12061511. PMID 32527022
- [Background] Han S, Choi JY. Prognostic value of 18F-FDG PET and PET/CT for assessment of treatment response to neoadjuvant chemotherapy in breast cancer: a systematic review and meta-analysis. Breast Cancer Res. 2020 Oct 31;22(1):119. doi: 10.1186/s13058-020-01350-2. PMID 33129348
- [Background] Wang Y, Zhang C, Liu J, Huang G. Is 18F-FDG PET accurate to predict neoadjuvant therapy response in breast cancer? A meta-analysis. Breast Cancer Res Treat. 2012 Jan;131(2):357-69. doi: 10.1007/s10549-011-1780-z. Epub 2011 Sep 30. PMID 21960111
- [Background] An YY, Kim SH, Kang BJ, Lee AW. Treatment Response Evaluation of Breast Cancer after Neoadjuvant Chemotherapy and Usefulness of the Imaging Parameters of MRI and PET/CT. J Korean Med Sci. 2015 Jun;30(6):808-15. doi: 10.3346/jkms.2015.30.6.808. Epub 2015 May 13. PMID 26028936
- [Background] Rouzier R, Perou CM, Symmans WF, Ibrahim N, Cristofanilli M, Anderson K, Hess KR, Stec J, Ayers M, Wagner P, Morandi P, Fan C, Rabiul I, Ross JS, Hortobagyi GN, Pusztai L. Breast cancer molecular subtypes respond differently to preoperative chemotherapy. Clin Cancer Res. 2005 Aug 15;11(16):5678-85. doi: 10.1158/1078-0432.CCR-04-2421. PMID 16115903